CLINICAL TRIAL: NCT05969080
Title: A Brief Intervention to Reduce Nonsuicidal Self-Injury and Improve Functioning in Veterans
Brief Title: Self-Injury Treatment and Recovery in Veterans
Acronym: STRIVe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4803-W; 1745432 (Other: VA IRB)
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Self-Injurious Behavior
Keywords: Self-Injurious Behavior; Veterans
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-SIB (Experimental): Participants randomized to the Treatment for Self-Injurious Behaviors (T-SIB) condition will receive nine sessions of T-SIB.
  Interventions: Behavioral: Treatment for Self-Injurious Behaviors
- Treatment As Usual (Active Comparator): Participants randomized to the TAU condition will be provided with referrals to both Durham VA and local community mental health resources and offered a consult for Durham VA mental health services.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Treatment for Self-Injurious Behaviors — Treatment for Self-Injurious Behaviors (T-SIB) incorporates evidence-based approaches to replace NSSI with behaviors that improve psychosocial functioning.
  Other Names: T-SIB
  Arms: T-SIB
Other: Treatment As Usual — Participants randomized to the TAU condition will be provided with referrals to both Durham VA and local community mental health resources and offered a consult for Durham VA mental health services.
  Other Names: TAU
  Arms: Treatment As Usual

SUMMARY:
Nonsuicidal self-injury (NSSI) refers to the intentional destruction of one's own body tissue without suicidal intent and for purposes that are not socially sanctioned. While NSSI has been understudied among Veterans, the lifetime prevalence rate of NSSI in Veterans is approximately three times higher than the general population. Moreover, NSSI is associated with increased risk for violence, psychiatric distress, and marked impairment in psychosocial functioning. Even though NSSI is distinct from suicidal behaviors in several important ways, NSSI remains a strong predictor of a future suicide attempt. The primary goal of this project is to evaluate the treatment and acceptability of a brief intervention for NSSI that aims to reduce psychosocial impairment and NSSI behaviors in Veterans.

DETAILED DESCRIPTION:
Nonsuicidal self-injury (NSSI) refers to the intentional destruction of one's own body tissue without suicidal intent and for purposes that are not socially sanctioned. While NSSI has been understudied among Veterans, the lifetime prevalence rate of NSSI in Veterans is approximately three times higher than the general population. Moreover, NSSI is associated with increased risk for violence, psychiatric distress, and marked impairment in psychosocial functioning. Even though NSSI is distinct from suicidal behaviors in several important ways, NSSI remains a strong predictor of a future suicide attempt. The primary goal of this project is to evaluate the treatment and acceptability of a brief intervention for NSSI that aims to reduce psychosocial impairment and NSSI behaviors in Veterans. This treatment, known as the Treatment for Self-Injurious Behaviors (T-SIB) incorporates evidence-based approaches to replace NSSI with behaviors that improve psychoso ial functioning. A core component of T-SIB is functional assessment that identifies the antecedents and consequences of NSSI. This project will enhance T-SIB by using ecological momentary assessment (EMA) to conduct NSSI functional assessment in-vivo. EMA reduces retrospective recall bias and can increase engagement with therapeutic goals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Past service in the United States military
* Nonsuicidal self-injury engagement on 2 occasions in past 30 days
* Fluent in English
* Able to provide voluntary informed consent

Exclusion Criteria:

* Lifetime history of psychosis, mania, or hypomania
* Imminent risk for suicide/homicide warranting immediate intervention
* Unable/unwilling to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by number of participants enrolled | 2 years after study enrollment begins
  All participants (N = 40) will need to be enrolled by the end of the second year of the study to consider the recruitment benchmark met.
Feasibility as measured rate of retention | End of treatment, about nine weeks after beginning the study
  Retention will be measured by the number of participants who complete at least six T-SIB treatment sessions. This benchmark will be considered meet if at least 2/3 of the 20 participants randomized to T-SIB complete at least 6 treatment sessions.

SECONDARY OUTCOMES:
Number of participants who report satisfaction with the T-SIB treatment | End of treatment, about nine weeks after beginning the study
  Participant satisfaction will be measured with the Client Satisfaction Questionnaire (CSQ-8). Total scores on the CSQ-8 range from 8 to 32, which higher scores indicating higher satisfaction. A cut score of 24 will be used such that if the CSQ-8 score exceeds 24, that patient is deemed to have been satisfied with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tate F Halverson, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No